CLINICAL TRIAL: NCT06468839
Title: The Impact of Addiction Management Model on Digital Addiction and Psychological Resilience in Second School Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Senem Celik Yavuz, phD student, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ANKARAUNIVERSITY-001
Record Dates: First submitted 2024-06-16; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Technology Addiction, Psychological Resilience, Risky Technology Use in Adolescent
Keywords: adolescent health, technology addiction, internet addiction health education, psychological resilience, emotional freedom tecnique.
MeSH Terms: conditions — Technology Addiction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): • Experimental group will receive the addiction management model. The addiction management model consists of a combination of standard education on addiction and emotional freedom techniques.
  They will receive 6 sessions of training:
  Weeks 1-4: Education on adolescence, addiction, and psychological resilience Weeks 5-6: Application of emotional freedom techniques.
  Interventions: Behavioral: digital addiction management model
- control (No Intervention): The control group receives only the standard education provided at the school.

INTERVENTIONS:
Behavioral: digital addiction management model — The experimental group will implement a digital addiction model. No intervention will be made to the control group.
  Arms: Experimental

SUMMARY:
Digital addiction has become a prevalent concern among adolescents, particularly middle school students. This study aims to develop and evaluate an addiction management model for 6th-grade students at risk of digital addiction. The model will combine standardized psychological resilience training with emotional freedom techniques to address both the behavioral and emotional aspects of digital addiction.

ELIGIBILITY:
Inclusion Criteria:

High risk of digital addiction as a result of the screening, Secondary school 6th grade students, Volunteering of the student and parent to participate in the research, The student must be able to speak, read and understand Turkish, The student does not have an auditory or mental disability that would affect his/her participation in the research.

Exclusion Criteria:

-

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2024-06-13 (Estimated); Study Completion 2024-06-13 (Estimated)

PRIMARY OUTCOMES:
Assessing Digital Addiction Risk Level | 1-3 month
  The Children and Adolescents' Digital Addiction Scale (CADAS) will be employed to evaluate the digital addiction risk level of the participants.• The CADAS scale ranges from 25 to 125, with higher scores indicating a greater risk of digital addiction.
  • A decrease in the scale score reflects a reduction in digital addiction risk

CONTACTS AND LOCATIONS:
Overall Officials: Ayfer TEZEL, professor, Study Chair — Ankara University
Locations (1):
- Senem Çelik Yavuz, Çankaya, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided